CLINICAL TRIAL: NCT00951041
Title: Safety and Immunogenicity Study of GSK Biologicals' Influenza Vaccine GSK2340272A in Adults Aged 18 to 60 Years
Brief Title: Study to Evaluate the Immunogenicity and Safety of an Investigational Influenza Vaccine (H1N1) in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 113574
Record Dates: First submitted 2009-07-31; First posted 2009-08-04 (Estimated); Results first posted 2018-11-26 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2017-04

CONDITIONS: Influenza
Keywords: influenza infection; GSK Bio's influenza vaccine GSK2340272A
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- GSK2340272A Group (Experimental): Healthy male or female adults, between and including 18 to 60 years of age, who received two doses of GSK2340272A vaccine. The first vaccine dose was administered intramuscularly in the deltoid region of the non-dominant arm at Day 0, and the second vaccine dose was administered intramuscularly in the deltoid region of the dominant arm at Day 21.
  Interventions: Biological: GSK investigational vaccine GSK2340272A
- GSK2340269A Group (Experimental): Healthy male or female adults, between and including 18 to 60 years of age, who received two doses of GSK2340269A vaccine. The first vaccine dose was administered intramuscularly in the deltoid region of the non-dominant arm at Day 0, and the second vaccine dose was administered intramuscularly in the deltoid region of the dominant arm at Day 21.
  Interventions: Biological: GSK investigational vaccine GSK2340269A

INTERVENTIONS:
Biological: GSK investigational vaccine GSK2340272A — Two intramuscular injections
  Arms: GSK2340272A Group
Biological: GSK investigational vaccine GSK2340269A — Two intramuscular injections
  Arms: GSK2340269A Group

SUMMARY:
The purpose of the study is to evaluate the safety and immunogenicity of GSK Biologicals' influenza vaccine GSK2340272A.

ELIGIBILITY:
Inclusion Criteria:

* A male or female aged 18 to 60 years at the time of the first vaccination.
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol
* Written informed consent obtained from the subject.
* Satisfactory baseline medical assessment by history and physical examination. Stable health status is defined as the absence of health event satisfying the definition of a serious adverse event, or a change in an ongoing drug therapy due to therapeutic failure or symptoms of drug toxicity, within one month prior to enrollment.
* Access to a consistent means of telephone contact, which may be either in the home or at the workplace, land line or mobile, but NOT a pay phone or multiple-user device.
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of the study vaccine or planned use during the study period.
* Presence of evidence of substance abuse or of neurological or psychiatric diagnoses which, although stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Presence of an axillary temperature ≥ 37.5°C, or acute symptoms greater than "mild" severity on the scheduled date of first vaccination. NOTE: The subject may be vaccinated at a later date, provided symptoms have resolved, vaccination occurs within the window specified by the protocol, and all other eligibility criteria continue to be satisfied.
* Diagnosed with cancer, or treatment for cancer, within the past 3 years.

  * Persons with a history of cancer who are disease-free without treatment for 3 years or more are eligible.
  * Persons with a history of histological-confirmed basal cell carcinoma of the skin successfully treated with local excisions only are excepted and may enroll within 3 years of diagnosis, but other histological types of skin cancer require a 3-year untreated and disease-free window as above.
  * Women who are disease free 3 years or more after the treatment for breast cancer and receiving long-term prophylactic are excepted and may enroll.
* Any confirmed or suspected immunosuppressive or immunodeficient condition including history of human immunodeficiency virus (HIV) infection.
* Clinically or virologically confirmed influenza infection within 6 months preceding the study start.
* Chronic administration of immunosuppressants or other immune modifying drugs within 6 months of study enrolment or planned administration during the study period.
* Receipt of any immunoglobulins and/or any blood products within 3 months of study enrolment or planned administration of any of these products during the study period.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin. Persons receiving individual doses of low molecular weight heparin outside of 24 hours prior to vaccination are eligible. Persons receiving prophylactic antiplatelet medications, e.g., low-dose aspirin, and without a clinically-apparent bleeding tendency, are eligible.
* An acute evolving neurological disorder or history of Guillain-Barré syndrome.
* Administration of any vaccines within 30 days before vaccination.
* Any known or suspected allergy to any constituent of influenza vaccines; a history of anaphylactic-type reaction to any constituent of influenza vaccines; or a history of severe adverse reaction to a previous influenza vaccine.
* Pregnant or lactating female
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Any conditions which, in the opinion of the investigator, prevents the subjects from participating in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2009-08-11 (Actual); Primary Completion 2010-08-30 (Actual); Study Completion 2010-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 113574 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113574 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113574 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113574 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113574 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113574 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113574 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GSK2340272A Group | GSK2340269A Group
Started | 64 | 66
Completed | 59 | 65
Not Completed | 5 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2340272A Group | GSK2340269A Group | Total
Number analyzed (Participants) | 64 | 66 | 130
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.90 (11.72) | 39.30 (13.16) | 39.60 (12.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 31 | 58
  Male | 37 | 35 | 72
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White-Caucasian/European heritage | 64 | 66 | 130

OUTCOME MEASURES:

1. Primary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against Flu A/California/7/2009 Strain of Influenza Disease
Description: Titers are presented as geometric mean titers (GMTs). The reference seropositivity cut-off value was equal to or above (≥) 1:10. The flu strain assessed was Flu A/California/7/2009 (H1N1)v-like, in subjects 18-60 years old. The primary endpoint results consist in those presented for GSK2340272A Group.
Time Frame: At Day 35
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects who received two doses of vaccine and for whom assay results were available for antibodies against H1N1 antigen for blood sample taken 14 days (Day 35) after the second vaccine dose.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 56 | 61
Titers | 780.2 [650.3 to 936.0] | 533.6 [412.2 to 690.7]

2. Primary Outcome: Number of Seroconverted Subjects for HI Antibodies
Description: Seroconversion (SCR) was defined as follows: for initially seronegative subjects, antibody titer equal to or above (≥) 1:40 after vaccination; for initially seropositive subjects, antibody titer after vaccination ≥ 4 fold the pre-vaccination antibody titer. The flu strain assessed was Flu A/California/7/2009 (H1N1)v-like, in subjects 18-60 years old. The primary endpoint results consist in those presented for GSK2340272A Group.
Time Frame: At Day 35
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects who received two doses of vaccine and for whom assay results were available for antibodies against H1N1 antigen for blood sample taken 14 days (Day 35) after the second vaccine dose.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 56 | 61
Participants | 56 | 60

3. Primary Outcome: Number of Seroprotected Subjects for HI Antibodies
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer equal to or above (≥) 1:40. The flu strain assessed was Flu A/California/7/2009 (H1N1)v-like, in subjects 18-60 years old. The primary endpoint results consist in those presented for GSK2340272A Group.
Time Frame: At Day 35
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 56 | 61
Participants | 56 | 61

4. Primary Outcome: Geometric Mean Fold Rise (GMFR) for HI Antibodies Against Flu A/California/7/2009 Strain of Influenza Disease
Description: GMFR, also called seroconversion factor (SCF), was defined as the fold increase in serum HI GMTs post-vaccination compared to pre-vaccination. The flu strain assessed was Flu A/California/7/2009 (H1N1)v-like, in subjects 18-60 years old. The primary endpoint results consist in those presented for GSK2340272A Group.
Time Frame: At Day 35
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 56 | 61
Fold change | 73.9 [55.1 to 99.2] | 45.6 [33.3 to 62.2]

5. Secondary Outcome: Titers for Serum HI Antibodies Against Flu A/California/7/2009 Strain of Influenza Disease
Description: Titers are presented as geometric mean titers (GMTs). The reference seropositivity cut-off value was equal to or above (≥) 1:10. The flu strain assessed was Flu A/California/7/2009 (H1N1)v-like, in subjects 18-60 years old.
Time Frame: At Days 0 and 21
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects who received two doses of vaccine and for whom assay results were available for antibodies against H1N1 antigen for blood samples taken at Day 0 and Day 21.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 56 | 61
Titers
  Flu A/California/7/2009, Day 0 | 10.6 [8.2 to 13.6] | 11.7 [8.7 to 15.8]
  Flu A/California/7/2009, Day 21 | 541.7 [415.7 to 706.0] | 530.5 [391.6 to 718.6]

6. Secondary Outcome: Titers for Serum HI Antibodies Against Flu A/California/7/2009 Strain of Influenza Disease
Description: as for outcome 5
Time Frame: At Day 182
Population: The analysis was performed on the ATP cohort for persistence (Month 6), which included all evaluable subjects who received at least one dose of the vaccine and for whom assay results were available for antibodies against H1N1 antigen for blood sample taken at Month 6.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 59 | 62
Titers | 161.9 [125.8 to 208.4] | 149.7 [109.9 to 203.8]

7. Secondary Outcome: Titers for Serum HI Antibodies Against Flu A/California/7/2009 Strain of Influenza Disease
Description: as for outcome 5
Time Frame: At Day 364
Population: The analysis was performed on the ATP cohort for persistence (Month 12), which included all evaluable subjects who received at least one dose of the vaccine and for whom assay results were available for antibodies against H1N1 antigen for blood sample taken at Month 12.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 58 | 63
Titers | 90.1 [68.9 to 117.8] | 96.0 [68.7 to 134.2]

8. Secondary Outcome: Number of Seroconverted Subjects for HI Antibodies
Description: Seroconversion (SCR) was defined as follows: for initially seronegative subjects, antibody titer equal to or above (≥) 1:40 after vaccination; for initially seropositive subjects, antibody titer after vaccination ≥ 4 fold the pre-vaccination antibody titer. The flu strain assessed was Flu A/California/7/2009 (H1N1)v-like, in subjects 18-60 years old.
Time Frame: At Day 21
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects who received two doses of vaccine and for whom assay results were available for antibodies against H1N1 antigen for blood sample taken at Day 21.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 56 | 61
Participants | 55 | 58

9. Secondary Outcome: Number of Seroconverted Subjects for HI Antibodies
Description: as for outcome 8
Time Frame: At Day 182
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 59 | 62
Participants | 53 | 49

10. Secondary Outcome: Number of Seroconverted Subjects for HI Antibodies
Description: as for outcome 8
Time Frame: At Day 364
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 58 | 63
Participants | 38 | 41

11. Secondary Outcome: Number of Seroprotected Subjects for HI Antibodies
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer equal to or above (≥) 1:40. The flu strain assessed was Flu A/California/7/2009 (H1N1)v-like, in subjects 18-60 years old.
Time Frame: At Days 0 and 21
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects who received two doses of vaccine and for whom assay results were available for antibodies against H1N1 antigen for blood sample taken at Day 0 and Day 21.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 56 | 61
Participants
  Flu A/California/7/2009, Day 0 | 7 | 8
  Flu A/California/7/2009, Day 21 | 55 | 60

12. Secondary Outcome: Number of Seroprotected Subjects for HI Antibodies
Description: as for outcome 11
Time Frame: At Day 182
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 59 | 62
Participants | 56 | 56

13. Secondary Outcome: Number of Seroprotected Subjects for HI Antibodies
Description: as for outcome 11
Time Frame: At Day 364
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 58 | 63
Participants | 48 | 51

14. Secondary Outcome: Seroconversion Factor (SCF) for HI Antibodies Against Flu A/California/7/2009 Strain of Influenza Disease
Description: SCF was defined as the fold increase in serum HI GMTs post-vaccination compared to pre-vaccination. The flu strain assessed was Flu A/California/7/2009 (H1N1)v-like, in subjects 18-60 years old.
Time Frame: At Day 21
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 56 | 61
Fold change | 51.3 [36.2 to 72.9] | 45.3 [32.6 to 63.0]

15. Secondary Outcome: SCF for HI Antibodies Against Flu A/California/7/2009 Strain of Influenza Disease
Description: as for outcome 14
Time Frame: At Day 35
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | GSK2340269A Group
Number analyzed (Participants) | 61
Fold change | 45.6 [33.3 to 62.2]

16. Secondary Outcome: SCF for HI Antibodies Against Flu A/California/7/2009 Strain of Influenza Disease
Description: as for outcome 14
Time Frame: At Day 182
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 59 | 62
Fold change | 15.3 [11.5 to 20.3] | 11.7 [8.7 to 15.9]

17. Secondary Outcome: SCF for HI Antibodies Against Flu A/California/7/2009 Strain of Influenza Disease
Description: as for outcome 14
Time Frame: At Day 364
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 58 | 63
Fold change | 8.4 [6.2 to 11.3] | 7.6 [5.6 to 10.4]

18. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) follow-up period after each dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects with the symptom sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 63 | 66
Participants
  Any Pain, Dose 1 | 56 | 39
  Grade 3 Pain, Dose 1 | 1 | 0
  Any Redness, Dose 1 | 20 | 3
  Grade 3 Redness, Dose 1 | 0 | 0
  Any Swelling, Dose 1 | 20 | 1
  Grade 3 Swelling, Dose 1 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 62 | 65
  Any Pain, Dose 2 | 53 | 33
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 62 | 65
  Grade 3 Pain, Dose 2 | 0 | 1
  Any Redness, Dose 2: number analyzed (Participants) | 62 | 65
  Any Redness, Dose 2 | 16 | 2
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 62 | 65
  Grade 3 Redness, Dose 2 | 0 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 62 | 65
  Any Swelling, Dose 2 | 12 | 1
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 62 | 65
  Grade 3 Swelling, Dose 2 | 0 | 0
  Any Pain, Across doses | 57 | 41
  Grade 3 Pain, Across doses | 1 | 1
  Any Redness, Across doses | 24 | 3
  Grade 3 Redness, Across doses | 0 | 0
  Any Swelling, Across doses | 21 | 2
  Grade 3 Swelling, Across doses | 0 | 0

19. Secondary Outcome: Number of Days With Solicited Local Symptoms
Description: The number of days with any solicited local symptoms reported during the solicited post-vaccination period.
Time Frame: During the 7-day (Days 0-6) follow-up period after each dose and overall
Population: The analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 64 | 66
Days
  Pain, Post-Dose 1 | 3.0 [3.0 to 5.0] | 2.0 [1.0 to 2.0]
  Pain, Post-Dose 2 | 3.0 [2.0 to 4.0] | 2.0 [1.0 to 2.0]
  Pain, Overall/dose | 3.0 [2.0 to 4.0] | 2.0 [1.0 to 2.0]
  Redness, Post-Dose 1 | 2.0 [1.0 to 3.5] | 4.0 [1.0 to 4.0]
  Redness, Post-Dose 2 | 2.0 [1.5 to 3.5] | 1.5 [1.0 to 2.0]
  Redness, Overall/dose | 2.0 [1.0 to 3.5] | 2.0 [1.0 to 4.0]
  Swelling, Post-Dose 1 | 3.0 [2.0 to 4.0] | 4.0 [4.0 to 4.0]
  Swelling, Post-Dose 2 | 3.0 [2.0 to 3.5] | 1.0 [1.0 to 1.0]
  Swelling, Overall/dose | 3.0 [2.0 to 4.0] | 2.5 [1.0 to 4.0]

20. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, headache, joint pain at other location, muscle aches, shivering, sweating and fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade and relationship to vaccination. Grade 3 symptom = symptom that prevented normal everyday activities. Grade 3 fever = fever above (>) 40.0 °C. Related = symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: During the 7-day (Days 0-6) follow-up period after each dose and across doses
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 63 | 66
Participants
  Any Fatigue, Dose 1 | 26 | 18
  Grade 3 Fatigue, Dose 1 | 2 | 1
  Related Fatigue, Dose 1 | 10 | 7
  Any Headache, Dose 1 | 19 | 10
  Grade 3 Headache, Dose 1 | 1 | 1
  Related Headache, Dose 1 | 9 | 5
  Any Joint Pain, Dose 1 | 15 | 5
  Grade 3 Joint Pain, Dose 1 | 1 | 0
  Related Joint Pain, Dose 1 | 9 | 2
  Any Muscle Aches, Dose 1 | 22 | 12
  Grade 3 Muscle Aches, Dose 1 | 1 | 0
  Related Muscle Aches, Dose 1 | 10 | 3
  Any Shivering, Dose 1 | 7 | 7
  Grade 3 Shivering, Dose 1 | 0 | 0
  Related Shivering, Dose 1 | 2 | 3
  Any Sweating, Dose 1 | 9 | 11
  Grade 3 Sweating, Dose 1 | 0 | 1
  Related Sweating, Dose 1 | 4 | 3
  Any Fever, Dose 1 | 1 | 0
  Grade 3 Fever, Dose 1 | 0 | 0
  Related Fever, Dose 1 | 1 | 0
  Any Fatigue, Dose 2: number analyzed (Participants) | 62 | 65
  Any Fatigue, Dose 2 | 29 | 13
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 62 | 65
  Grade 3 Fatigue, Dose 2 | 3 | 0
  Related Fatigue, Dose 2: number analyzed (Participants) | 62 | 65
  Related Fatigue, Dose 2 | 16 | 7
  Any Headache, Dose 2: number analyzed (Participants) | 62 | 65
  Any Headache, Dose 2 | 19 | 12
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 62 | 65
  Grade 3 Headache, Dose 2 | 3 | 0
  Related Headache, Dose 2: number analyzed (Participants) | 62 | 65
  Related Headache, Dose 2 | 11 | 5
  Any Joint Pain, Dose 2: number analyzed (Participants) | 62 | 65
  Any Joint Pain, Dose 2 | 23 | 7
  Grade 3 Joint Pain, Dose 2: number analyzed (Participants) | 62 | 65
  Grade 3 Joint Pain, Dose 2 | 2 | 1
  Related Joint Pain, Dose 2: number analyzed (Participants) | 62 | 65
  Related Joint Pain, Dose 2 | 15 | 3
  Any Muscle Aches, Dose 2: number analyzed (Participants) | 62 | 65
  Any Muscle Aches, Dose 2 | 30 | 7
  Grade 3 Muscle Aches, Dose 2: number analyzed (Participants) | 62 | 65
  Grade 3 Muscle Aches, Dose 2 | 2 | 0
  Related Muscle Aches, Dose 2: number analyzed (Participants) | 62 | 65
  Related Muscle Aches, Dose 2 | 17 | 2
  Any Shivering, Dose 2: number analyzed (Participants) | 62 | 65
  Any Shivering, Dose 2 | 12 | 4
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 62 | 65
  Grade 3 Shivering, Dose 2 | 1 | 0
  Related Shivering, Dose 2: number analyzed (Participants) | 62 | 65
  Related Shivering, Dose 2 | 10 | 2
  Any Sweating, Dose 2: number analyzed (Participants) | 62 | 65
  Any Sweating, Dose 2 | 12 | 7
  Grade 3 Sweating, Dose 2: number analyzed (Participants) | 62 | 65
  Grade 3 Sweating, Dose 2 | 1 | 0
  Related Sweating, Dose 2: number analyzed (Participants) | 62 | 65
  Related Sweating, Dose 2 | 8 | 1
  Any Fever, Dose 2: number analyzed (Participants) | 62 | 65
  Any Fever, Dose 2 | 2 | 0
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 62 | 65
  Grade 3 Fever, Dose 2 | 0 | 0
  Related Fever, Dose 2: number analyzed (Participants) | 62 | 65
  Related Fever, Dose 2 | 1 | 0
  Any Fatigue, Across doses | 35 | 23
  Grade 3 Fatigue, Across doses | 5 | 1
  Related Fatigue, Across doses | 20 | 11
  Any Headache, Across doses | 30 | 18
  Grade 3 Headache, Across doses | 4 | 1
  Related Headache, Across doses | 17 | 8
  Any Joint Pain, Across doses | 27 | 10
  Grade 3 Joint Pain, Across doses | 2 | 1
  Related Joint Pain, Across doses | 18 | 5
  Any Muscle Aches, Across doses | 35 | 14
  Grade 3 Muscle Aches, Across doses | 2 | 0
  Related Muscle Aches, Across doses | 18 | 5
  Any Shivering, Across doses | 16 | 10
  Grade 3 Shivering, Across doses | 1 | 0
  Related Shivering, Across doses | 10 | 4
  Any Sweating, Across doses | 17 | 14
  Grade 3 Sweating, Across doses | 1 | 1
  Related Sweating, Across doses | 11 | 4
  Any Fever, Across doses | 3 | 0
  Grade 3 Fever, Across doses | 0 | 0
  Related Fever, Across doses | 2 | 0

21. Secondary Outcome: Number of Days With Solicited General Symptoms
Description: The number of days with any solicited general symptoms reported during the solicited post-vaccination period.
Time Frame: During the 7-day (Days 0-6) follow-up period after each dose and overall
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 64 | 66
Days
  Fatigue, post-Dose 1 | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0]
  Fatigue, post-Dose 2 | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0]
  Fatigue, Overall/dose | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0]
  Headache, post-Dose 1 | 2.0 [1.0 to 3.0] | 1.5 [1.0 to 2.0]
  Headache, post-Dose 2 | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0]
  Headache, Overall/dose | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 2.0]
  Joint pain, post-Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [2.0 to 3.0]
  Joint pain, post-Dose 2 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Joint pain, Overall/dose | 2.0 [1.0 to 3.0] | 2.0 [1.5 to 3.0]
  Muscle aches, post-Dose 1 | 2.0 [1.0 to 3.0] | 1.5 [1.0 to 2.0]
  Muscle aches, post-Dose 2 | 2.0 [2.0 to 3.0] | 3.0 [1.0 to 3.0]
  Muscle aches, Overall/dose | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Sweating, post-Dose 1 | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0]
  Sweating, post-Dose 2 | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0]
  Sweating, Overall/dose | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0]
  Shivering, post-Dose 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 2.0]
  Shivering, post-Dose 2 | 1.0 [1.0 to 2.0] | 2.0 [1.5 to 2.0]
  Shivering, Overall/dose | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Fever, post-Dose 1 | NA [NA to NA] — This symptom was not reported for the first dose of study vaccine. | NA [NA to NA] — This symptom was not reported for GSK2340269A Group.
  Fever, post-Dose 2 | 1.0 [1.0 to 1.0] | NA [NA to NA] — This symptom was not reported for GSK2340269A Group.
  Fever, Overall/dose | 1.0 [1.0 to 1.0] | NA [NA to NA] — This symptom was not reported for GSK2340269A Group.

22. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During the 21-day (Days 0-20) follow-up after the first vaccination and during the 63-day (Days 21-83) follow-up after the second vaccination (From Day 0 to Day 84)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 64 | 66
Participants
  Any AE(s) | 22 | 27
  Grade 3 AE(s) | 1 | 4
  Related AE(s) | 5 | 6

23. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (From Day 0 up to Day 364)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 64 | 66
Participants | 0 | 3

24. Secondary Outcome: Number of Subjects With Adverse Events of Specific Interest (AESI)
Description: An AESI was defined as an AE including autoimmune diseases and other mediated inflammatory disorders and assessed by the investigator as specific to the treatment administration.
Time Frame: During the entire study period (From Day 0 up to Day 364)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group | GSK2340269A Group
Number analyzed (Participants) | 64 | 66
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) post-vaccination period. Unsolicited AEs: from Day 0 to Day 84. SAEs: during the entire study period (from Day 0 up to Day 364).
Description: Solicited local and general symptoms were collected only from subjects with their symptom sheet completed.
Arm/Group | GSK2340272A Group | GSK2340269A Group
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/64 | 3/66
Other Adverse Events (participants affected / at risk) | 61/64 | 49/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2340272A Group (N=64) | GSK2340269A Group (N=66)
Hypersensitivity (Immune system disorders) | 0 | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | GSK2340272A Group (N=64) | GSK2340269A Group (N=66)
Nasopharyngitis (Infections and infestations) | 5 | 4
Influenza like illness (General disorders) | 1 | 6
Pain (General disorders) | 57/63 | 41 — This solicited local symptom was only collected from subjects with their symptom sheet completed.
Redness (General disorders) | 24/63 | 3 — This solicited local symptom was only collected from subjects with their symptom sheet completed.
Swelling (General disorders) | 21/63 | 2 — This solicited local symptom was only collected from subjects with their symptom sheet completed.
Fatigue (General disorders) | 35/63 | 23 — This solicited general symptom was only collected from subjects with their symptom sheet completed.
Headache (General disorders) | 30/63 | 18 — This solicited general symptom was only collected from subjects with their symptom sheet completed.
Joint pain (General disorders) | 27/63 | 10 — This solicited general symptom was only collected from subjects with their symptom sheet completed.
Muscle aches (General disorders) | 35/63 | 14 — This solicited general symptom was only collected from subjects with their symptom sheet completed.
Shivering (General disorders) | 16/63 | 10 — This solicited general symptom was only collected from subjects with their symptom sheet completed.
Sweating (General disorders) | 17/63 | 14 — This solicited general symptom was only collected from subjects with their symptom sheet completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.